CLINICAL TRIAL: NCT02421016
Title: A Prospective, Randomized Trial of SYNERGY Bioresorbable Polymer Coated Stents Versus ABSORB Bioresorbable Backbone Stents in Patients Undergoing Coronary Stenting (ISAR-RESORB)
Brief Title: Test Efficacy With Bioresorbable Polymer Coating Versus Bioresorbable Polymer Backbone (ISAR-RESORB)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No S03914
Record Dates: First submitted 2015-04-09; First posted 2015-04-20 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Stenosis
Keywords: De novo stenosis; bioresorbable polymer coating; bioresorbable polymer backbone
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SYNERGY EES (Experimental): Bioresorbable polymer everolimus-eluting stent
  Interventions: Device: SYNERGY EES
- ABSORB [BVS] (Active Comparator): Everolimus-eluting bioresorbable backbone stent
  Interventions: Device: ABSORB [BVS]

INTERVENTIONS:
Device: SYNERGY EES — Bioresorbable polymer everolimus-eluting stent
  Arms: SYNERGY EES
Device: ABSORB [BVS] — Everolimus-eluting bioresorbable backbone stent
  Arms: ABSORB [BVS]

SUMMARY:
The bioresorbable polymer SYNERGY EES exhibits a favourable vascular healing profile in patients undergoing coronary intervention for de novo lesions. Specifically, the SYNERGY EES is superior to the ABSORB bioresorbable vascular scaffold in terms of antirestenotic efficacy as assessed by angiography at 6-8 months.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) with drug-eluting stent (DES) implantation currently represents the dominant treatment strategy in patients undergoing catheter intervention. However, effective neointimal suppression occurs at the cost of a systematic delay in arterial healing in comparison with after bare metal stenting. This underlies a small but significant increased risk of stent thrombosis after DES implantation in comparison with bare metal stent implantation as well as a possible excess of in-stent neoatheroma formation. To address this issue recent technological advances have focused on bioresorbable polymer coatings and the development of stents with fully resorbable backbones.

Newer generation metallic DES with bioresorbable polymer coatings have been shown to improve vascular healing after coronary stenting. In particular a novel thin-strut bioresorbable polymer everolimus-eluting stent (EES, SYNERGY, Boston Scientific Corp., Natick, MA, USA) has shown high angiographic antirestenotic efficacy as well as high clinical efficacy and safety in early randomized trials. In addition, DES with bioresorbable backbones represent an alternative approach to ensure short-term vessel scaffolding and drug delivery with enhanced vessel healing. The everolimus-eluting bioresorbable backbone stent (ABSORB bioresorbable vascular scaffold [BVS], Abbott Vascular, Santa Rosa, CA, USA) is the most-extensively studied device in this class and early reports in selected patients show encouraging clinical results. However requirement for thicker stent struts and more careful lesion preparation has led to concerns that potential clinical benefits may be offset by erosion of early antirestenotic efficacy and occurrence of clinical events related to limitations of device deployment.

At present there is a lack of randomized clinical trial data examining outcomes of patients treated with these two alternative strategies. The aim of the current ISAR-RESORB study is to test the clinical performance of the bioresorbable-polymer SYNERGY with that of the ABSORB BVS in patients undergoing PCI of de novo coronary lesions. The primary endpoint will be percentage diameter stenosis at protocol-mandated 6-8 month angiographic follow-up. Secondary clinical endpoint will be assessed at 12 months. Sample size calculation is based on a superiority hypothesis for SYNERGY versus ABSORB BVS. It is planned to enrol a total of 230 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with ischemic symptoms or evidence of myocardial ischemia in the presence of ≥ 50% de novo stenosis located in native coronary vessels (max. 2 lesions in 2 separate vessels)
* Reference diameter ≥2.5 mm and ≤3.9 mm
* Lesion length <28 mm
* Written, informed consent by the patient for participation in the study

Exclusion Criteria:

* Cardiogenic shock
* Acute ST-elevation myocardial infarction within 48 hours from symptom onset.
* Target lesion located in left main trunk or bypass graft
* Severe calcification of the lesion
* Target lesion contains a side branch (diameter ≥2mm) or a bifurcation or is located 2 mm away from a bifurcation
* Ostial lesions
* Severe vessel tortuosity
* Renal insufficiency (most recent serum creatinine within the last 72h prior to randomization > 2 mg/dl or 177 µmol/l)
* Malignancies or other co-morbid conditions with life expectancy less than 12 months or that may result in protocol non-compliance
* Pregnancy, present (positive pregnancy test), suspected or planned, breast feeding
* Contraindications or allergy to platinum, chromium, everolimus or the inability to take antiplatelet therapy for at least 6 months after stenting; known allergy to PLLA, PDLLA or PLGA polymer
* Previous enrollment in this trial
* Patient's inability to fully cooperate with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Percentage diameter stenosis (in-stent) by quantitative coronary angiography analysis | at 6-8 months

SECONDARY OUTCOMES:
Composite of cardiac death/target vessel-myocardial infarction (MI)/ target lesion revascularization (TLR) (Device-oriented composite endpoint) | at 12 months
Composite of death/any MI/all revascularization (Patient-oriented composite endpoint) | at 12 months
Composite of cardiovascular death or MI | at 12 months
Stent Thrombosis | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Byrne, MB BCh PhD, Principal Investigator — Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum München, Munich, Bavaria, Germany